CLINICAL TRIAL: NCT02349945
Title: Significance of the FSH Receptor Polymorphism p.N680S for the Efficacy of FSH Therapy of Idiopathic Male Infertility: a Pharmacogenetic Approach
Brief Title: FSH Receptor Polymorphism p.N680S and Efficacy of FSH Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Collaborators: University of Roma La Sapienza (Other); University of Halle Medical Faculty (Other); Istituto Clinico Humanitas (Other); University of Padova (Other); University of Florence (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Professor, Azienda USL Modena
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2010-020240-35
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): FSHR A680G SNP homozygous for allele N treated with follitropin alpha
  Interventions: Drug: follitropin alpha
- Arm 2 (Experimental): FSHR A680G SNP homozygous for allele S treated with follitropin alpha
  Interventions: Drug: follitropin alpha

INTERVENTIONS:
Drug: follitropin alpha — All subjects included in the study will receive recombinant FSH therapy (follitropin alpha: Gonal-f 150 I.U. s.c. every other day for 12 weeks). Follow up: 12 further weeks after end of treatment.
  Previous studies included in the Cochrane meta-analysis used: hMG/hCG, 150 IU three times a week for 13 weeks; purified FSH, 150 IU/day for 12 weeks; rec hFSH, 150 IU/day for 12 weeks; rec hFSH, 100 IU on alternate days for 3 months. Therefore any dosage > 100 IU on alternate days is eligible. The duration of treatment is based on the duration of one spermatogenetic cycle.
  Other Names: Gonal f

SUMMARY:
CONDITION: Idiopathic male infertility In men with idiopathic infertility, the sperm DNA fragmentation index (DFI) within 12 weeks of FSH therapy and 12 weeks follow-up improves depending on the FSHR genotype as assessed by the non-synonymous SNP rs6166 (wild type or p.N680S).

This is a phase II b, multicenter, prospective, open label, one arm, clinical trial stratified according to the patient's genotype.

INTERVENTION: FSH therapy (150 I.U. sc every other day for 12 weeks) in infertile men who are homozygous for the wild-type FSHR or the p.N680S allele of the FSHR. Duration of intervention per patient: 12 weeks

Primary efficacy endpoint: Sperm DFI. Number of patients with an improvement in DFI > 60% Key secondary endpoint(s): pregnancy, semen parameters, serum levels of inhibin B and AMH.

DETAILED DESCRIPTION:
Male factor infertility is responsible for about 50% of cases of involuntary couple infertility and remains idiopathic in about half of the cases. At present, there are no consistently effective treatments for male idiopathic infertility. Since follicle-stimulating hormone (FSH) is fundamental for spermatogenesis, recombinant hFSH is empirically used for male infertility treatment. The response to FSH, however, is highly variable and while sperm parameters improve in some patients, about 50% of the subjects do not clearly respond to FSH. Several studies were performed in the past and a recent Cochrane meta-analysis showed that FSH treatment of male idiopathic infertility overall significantly improves pregnancy rate. Nevertheless, no predictive marker of response to FSH, allowing a stratified therapeutic approach, was identified so far.

The sperm DNA fragmentation index (DFI) provides an estimation of genetic integrity of spermatozoa and was shown to improve significantly after FSH treatment. Therefore, DFI could be used as a pharmacodynamic marker of FSH in the male.

In women, the response to FSH varies depending on the FSH receptor (FSHR) genotype, as determined by the non-synonymous SNP rs6166, which exchanges the amino acid Asn to Ser in codon 680. This SNP is very common, with a minor allele frequency of 0.4. Women homozygous for Ser at amino acid position 680 of the FSHR are less sensitive to endogenous and exogenous FSH compared to those homozygous for Asn and require more FSH for multiple follicular growth and maturation in assisted reproduction. The investigators hypothesize that the variable response to FSH in unselected infertile men is due to a different individual sensitivity to FSH as determined by the common FSHR polymorphism rs6166. In particular the investigators will test the hypothesis that men homozygous for Asn at 680 (wild type) will respond better to exogenous FSH treatment in terms of sperm DFI compared to men homozygous for Ser, assessing sperm DFI as pharmacodynamic parameter of FSH.

Men with idiopathic infertility and normal serum FSH levels, candidate for treatment with FSH, will be recruited. Men with a sperm DFI > 15% will be included in the trial if carriers of the homozygous Asn/Asn or Ser/Ser at aminoacid position 680. The FSHR genotype will be assessed centrally and the physician will only receive the information whether the patient is eligible for entering the trial (i.e. homozygous) but both the physician and the patient will remain blind to the genotype. Human recombinant FSH (Gonal-f, Merck Serono) will be self-administered sc at the dose of 150 IU every other day for 12 weeks, followed by 12 weeks of observation (follow up). Changes in sperm DFI will be the primary end point and compared between the two arms. In addition, the effects on pregnancy rate and other clinical and hormonal parameters will be evaluated.

Should this pilot, proof-of-principle trial demonstrate that the response to FSH in male idiopathic infertility depends on FSHR genotype, larger interventional trials aiming at assessing the effects on pregnancy rate will be justified.

ELIGIBILITY:
Inclusion Criteria:

* age 20-50 years
* idiopathic male factor infertility for at least one year;
* homozygous FSHR allele at codon 680 (wild type: Asn/Asn or Ser/Ser);
* sperm DFI > 15%;
* normal serum FSH levels (< 8 IU/L)
* normal serum LH, testosterone, prolactin and estradiol levels
* normal ovulatory female partner These men might have impaired ejaculate parameters (decreased sperm count and/or decreased proportion of sperm with progressive motility and/or decreased proportion of sperm with normal morphology) of unknown aetiology.

Exclusion Criteria:

* azoospermia
* all known aetiologies of male infertility (endocrine disorders, genetic disorders, chromosome abnormalities, congenital bilateral absence of the vas deferens, microdeletions within the AZF regions of the Y chromosome, varicocele, cryptorchidism, infections, immunological infertility, and obstructive infertility)
* all known aetiologies of female infertility in the partner (tubal blockage, endocrine abnormalities including anovulation and PCO, anatomical abnormalities, infections)
* heterozygous FSHR allele at codon 680
* drug abuse and major systemic diseases
* testicular insufficiency

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sperm DFI | "after 12 weeks"

SECONDARY OUTCOMES:
Sperm DFI (DNA Fragmentation Index) | "Baseline"
Sperm DFI | "after 24 weeks"

OTHER OUTCOMES:
Pregnancy rate | "baseline"
Pregnancy rate | "After 12 weeks"
Pregnancy rate | "after 24 weeks"
Sperm count | "baseline"
Sperm count | "after 12 weeks"
Sperm count | "after 24 weeks
Inhibin B | "baseline"
  Serum dosage
Inhibin B | "after 12 weeks"
  Serum dosage
Inhibin B | "after 24 weeks"
  Serum dosage
Anti-Mullerian Hormone (AMH) | "baseline"
  Serum dosage of Anti-Mullerian Hormone
AMH | "after 12 weeks"
  Serum dosage of Anti-Mullerian Hormone
AMH | "after 24 weeks"
  Serum dosage of Anti-Mullerian Hormone

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Simoni, MD, PhD, Principal Investigator — Azienda USL Modena
Locations (6):
- Zentrums für Reproduktions-medizin und Andrologie Universitätsklinikum Halle (Saale), Martin-Luther-Universität Halle-Wittenberg, Halle, Germany
- Italy (5):
  - Dipartimento di Ginecologia e Medicina della Riproduzione IRCCS Istituto Clinico Humanitas,, Rozzano, Milan
  - Andrology Unit Department of Clinical Physiopathology, Florence
  - AziendaUSLModena, Modena
  - University of Padova Department of Histology, Microbiology and Medical Biotechnologies Clinical Pathology Section & Centre for Male Gamete Cryopreservation, Padua
  - Department of Medical Pathophysiology, University of Rome La Sapienza, Lab of Seminology & Immunology of Reproduction, Rome